CLINICAL TRIAL: NCT06746584
Title: Investigation of the Effect of Benson Relaxation Exercise on Anxiety and Sleep Quality in Inpatients in Psychiatric Service: a Randomized Controlled Study
Brief Title: Benson Relaxation Exercise on Anxiety and Sleep Quality in Psychiatric Service (BREASQPS)
Acronym: (BREASQPS)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, elçin babaoğlu, Asst. Dr. (Psychiatric Nursing), Uskudar University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 61351342/020-391
Record Dates: First submitted 2024-11-29; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Sleep Quality; Anxiety
Keywords: psychiatric inpatients, Benson relaxation, sleep Quality, anxiety
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: randomized controlled trial single blinded
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Since patients diagnosed with psychotic disorder and schizophrenia have delusions and hallucinations, the effect of some instructions in the Benson relaxation technique on these symptoms cannot be known. Therefore, it was planned to exclude psychosis and schizophrenia patients with delusions and hallucinations from the study.
  Interventions: Behavioral: benson relaxation exercise
- Control Group (No Intervention): Since patients diagnosed with psychotic disorder and schizophrenia have delusions and hallucinations, the effect of some instructions in the Benson relaxation technique on these symptoms cannot be known. Therefore, it was planned to exclude psychosis and schizophrenia patients with delusions and hallucinations from the study

INTERVENTIONS:
Behavioral: benson relaxation exercise — BRT is one of the behavioural intervention techniques developed by Herbert Benson in 1975. BRT is based on the principle of deep breathing and relaxing all the muscles in the body by choosing a word that is meaningful for the individual and focusing on it. This exercise, which has no side effects on patients and can be applied for patients of all age groups, is more widely used because it is a simple and easy-to-learn method compared to other relaxation methods all the muscles in the body by choosing a word that is meaningful for the individual and focusing on it.
  Other Names: benson relaxation
  Arms: Intervention Group

SUMMARY:
This study was planned to investigate the effect of Benson Relaxation Exercise on anxiety and sleep quality in inpatients in psychiatric ward. The following hypothesis will be tested in the study.

H1: Anxiety level of the patients who underwent Benson relaxation exercise is lower than the patients who did not undergo Benson relaxation exercise.

H2: The sleep quality of patients who undergo Benson relaxation exercise is better than patients who do not undergo Benson relaxation exercise.

The study is designed as a single-blind, randomised controlled trial. The study will be conducted in four psychiatric wards of a private psychiatric hospital in Turkey between 18.11.2024-06.06.2025. Verbal and written informed consent will be obtained from participants or their legal guardians before assignment to study groups. The study will be conducted according to the CONSORT flow diagram (http://www.consort-statement.org/consort-statement/flow-diagram) (2010)

DETAILED DESCRIPTION:
The study will be conducted between 18.11.2024 and 06.06.2025 in four psychiatric wards of a private psychiatric hospital in Turkey. In this hospital, patients with schizophrenia, psychotic disorders, mood and anxiety disorders and substance use disorders receive inpatient treatment. In the last 1 year, a total of 350 patients received inpatient treatment in the hospital. Patients stay in single rooms in the clinics. Apart from medical treatment and care, patients participate in activities such as group activities, occupational hours and walking.

Participants The population of this study consisted of a total of 350 inpatients in psychiatric wards. Since patients diagnosed with psychotic disorder and schizophrenia have delusions and hallucinations, the effect of some instructions in the Benson relaxation technique on these symptoms cannot be known. Therefore, it was planned to exclude psychosis and schizophrenia patients with delusions and hallucinations from the study. In sample selection, State Anxiety Form I (STAI-I) / State Anxiety Form II (STAI-I) and Pittsburg Sleep Quality Index (PSQI) will be applied by the researchers to patients other than these diagnoses. In the literature, the mean score of the STAI I-II scale varies between 36 and 41. Scores between 20 and 39 indicate mild anxiety and 40-59 points indicate moderate anxiety . In the literature, PSQI total score has a value between 0-21. A total scale score of 5 and above indicates poor sleep quality. Since the differences in anxiety and sleep quality levels will affect group homogeneity, patients with a total score of 20-59 points (mild and moderate) from STAI-I-II and patients with a score above 5 from PSQI will constitute the sample of the study. Accordingly, the inclusion criteria were planned as follows: Patients aged 18 years and over, patients being treated for mood, anxiety, obsessive-compulsive disorder and substance use disorder, patients with STAI I-II scores between 20 and 59, patients with PSQI score above 5. Exclusion criteria were patients under 18 years of age, patients with psychotic disorders with hallucinations and delusions, patients with schizophrenia, STAI I-II score below 20 and above 59, PSQI score below 5. Patients who meet the inclusion criteria will be divided into two groups as intervention and control group by single blind randomisation. In the randomisation phase of the study, Statistical Analysis Software will be used to randomly assign patients. Patients will be randomly assigned to groups using this programme. Patients included in the study will be numbered according to the order of arrival and placed in the intervention and control groups according to the order in the randomisation list.

It is planned that one of the researchers will assign the patients to the groups using the Statistical Analysis Software programme. This investigator will not participate in the Benson exercises with the patients. Since none of the investigators knew which patients participated in the study group, the study was conducted using single blinding method.

Accordingly, it is planned to finalise the study when a total of 70 patients, 35 in the intervention group and 35 in the control group, are reached. After reaching a sample of 70 people, it is planned to perform the power analysis of the study with GPower 3.1 programme at 95% confidence interval.

Measurement In this study, the patient descriptive information form, STAI-II and PSQI forms created by the researchers will be used. Patient Descriptive Information Form: This form developed by the researchers includes 8 number of questions to determine sociodemographic characteristics such as age, gender, educational status, duration of illness, number of hospitalisations, family history of illness, age at onset of illness and psychotropic drugs used. The State-Trait Anxiety Inventory Anxiety (STAI I-II): This scale was developed by Spielberger et.al. (1983) and its Turkish validity and reliability was performed by Öner and Le Compte (1983). The scale measures anxiety in both healthy and clinical populations. The scale consists of two parts: State Anxiety Inventory (STAI I) and Trait Anxiety Inventory (STAI II). STAI I determines how the individual feels at a certain time and under certain conditions, while STAI II determines how the individual feels regardless of the situation and conditions in which the individual is located. Alpha reliability coefficient of the scale was determined between 0.94-0.96 for STAI I and 0.83-0.87 for STAI II. Each scale consists of two types of statements with 20 items. Direct statements describe negative emotions and inverted statements describe positive emotions. The reversed statements are items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20 in STAI I and items 21, 26, 27, 30, 33, 36 and 39 in STAI II. In STAI I, the answers were evaluated with a 4-point scale (not at all, a little, a lot, completely). In STAI II, participants' responses were measured with a 4-point scale (never, sometimes, very often, almost always). The total score value obtained from both scales is between 20 and 80. It has also been shown that people with higher scores on the STAI scales are more prone to experience anxiety. The scale has been translated into 48 languages as of 2011. The STAI I AND II have been shown to have excellent psychometric properties with good reliability and validity. Pittsburgh Sleep Quality Index -PSQI (The Pittsburgh Sleep Quality Index): The Turkish validity and reliability of this scale developed by Buysse et al. (1989) was performed by Ağargün et al. (1996) The PSQI provides a quantitative measure of sleep quality that helps to define good and bad sleep. The PSQI contains a total of 24 questions. 19 of these questions are self-assessment questions. 5 questions are answered by the individual's spouse or a friend. These 5 questions are used only for clinical information and do not participate in the evaluation. Question 19 of the self-assessment questions is related to the presence of a roommate or spouse and is not taken into account in determining the total and component scores of the scale. Self-assessment questions include various factors related to sleep quality. These questions determine sleep duration, sleep latency, and the frequency and severity of special problems related to sleep. The 18 scored items were grouped into 7 component scores. Some of the components consist of a single item, while others are obtained by grouping several items. Each item is evaluated with a score between 0-3. The sum of the seven component scores gives the total PSQI score. The total score has a value between 0-21. A high total scale score indicates poor sleep quality. A total PSQI score of 5 and above indicates poor sleep quality. Data collection tools will be applied to both intervention and control groups by the researchers before starting BRT. At the end of 2 weeks, immediately after the completion of all exercises, final measurements will be made with the same data collection tools to both groups. At the end of 2 weeks, after the Benson exercises are completed, follow-up measurements will be performed with the same measurement tools in both groups for follow-up evaluation in the 3rd week. While BRT is applied to the intervention group, no application will be made to the patients in the control group. Measurement tools will be applied to the control group at the same time intervals as the patients in the intervention group.

Prosedur In the study, it is planned to use training booklets containing Benson application steps to be given to the intervention group. The content of the training booklets will be created by the researchers and expert opinion will be obtained from a psychiatrist, a psychologist and a psychiatric nurse about its application in psychiatry clinics. After the expert opinion, it is planned to carry out a pre-application with 6 patients who meet the research criteria and agree to participate in the study in order to obtain the comprehensibility of the commands in both the data collection forms and this booklet, the adequacy of the duration and the feedback of the patients. After the preliminary application, it is planned to make the necessary changes in the data collection forms and training booklets. BRT is one of the behavioural intervention techniques developed by Herbert Benson in 1975. BRT is based on the principle of deep breathing and relaxing all the muscles in the body by choosing a word that is meaningful for the individual and focusing on it. This exercise, which has no side effects on patients and can be applied for patients of all age groups, is more widely used because it is a simple and easy-to-learn method compared to other relaxation methods. Below are the stages of the Benson relaxation exercise. These stages are given as commands to the person doing the exercise by the practitioner in the form of commands. The exercise lasts between 10 and 20 minutes on average. The commands to be given to the intervention group in the application phase of the research are as follows. 1. Choose a short sentence or a word that is meaningful for you and that you can concentrate your attention on. This can be 'health, prosperity, abundance' or 'love'. 2. Sit quietly in a comfortable position. 3. Close your eyes. 4. Relax the muscles in your calves, thighs, abdomen, chest, shoulders, shoulders, neck and head, starting from your feet and gradually moving upwards towards your upper muscle groups. 5. Breathe slowly and naturally and say your focus word, sound, phrase or prayer silently to yourself as you exhale. 6. Maintain a passive attitude. Do not worry about whether you are doing well or not. When other thoughts come to mind, simply say to yourself, 'Everything is good', 'I am light, healthy and fit' and calmly focus on your breathing and muscles. 7.Focus on relaxation, on relaxation until the commands are finished. 8.Do not stand up immediately after the commands are finished. Continue to sit quietly for a minute or two so that you can return to the environment you are in. Then open the tapes on your eyes, slowly open your eyes and sit for another minute or two before getting up. Intervention Phase Although the length of hospital stay of the patients in this study varies depending on their mental status and treatment progress, as a standard practice of the hospital, patients are treated in the clinic for an average of three weeks in the hospital. For this reason, it is planned to apply BRT to the intervention group for 2 weeks and to make a follow-up evaluation in the 3rd week. This exercise, which will be applied to the patients in the intervention group through individual sessions once a day for two weeks during their hospital stay, is planned to be performed in a quiet room with each session lasting 20 minutes. BRT will be applied to the intervention group by a psychiatric nurse trained in exercises in an environment supervised by the researchers. The application is planned to be carried out in the afternoon in a quiet environment with few environmental stimuli. The exercises are planned to be applied individually to each patient. In the application, the psychiatric nurse will give commands to the patient about relaxation techniques. After the first application, the nurse will stay with the patient until the end of the application to reduce possible problems that may arise from sudden changes in the patient's condition and to ensure that the patient successfully completes the relaxation exercise process. Patients in the control group will continue to receive standard treatment and care at the hospital. No other intervention was made to the control group during the study. All participants in the intervention and control groups will continue to receive combinations of medication and psychotherapy.

Statistical analysis of the data

Statistical analyses will be performed using the Statistical Package for the Social Sciences (SPSS v26.0, IBM Corp., Armonk, NY, USA). Descriptive data will be presented as mean, frequency, percentage and standard deviation. Chi-square and Fisher's tests will be used to assess differences in qualitative characteristics (e.g. gender, education, marital status) between the two groups. Furthermore, independent sample t-tests are planned to be used to examine differences in mean scores between the intervention and control groups (e.g. STAI I-II, Pittsburg Sleep). Analysis of covariance (ANCOVA) is planned to compare anxiety and sleep quality scores between the intervention and control groups in the post-intervention post-test, controlling for confounding variables (e.g. pre-test score and group factors). A significance level of 0.05 will be applied for all statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over,
* patients being treated for mood, anxiety, obsessive-compulsive disorder and substance use disorder,
* patients with STAI I-II scores between 20 and 59, patients with PSQI score above 5.

Exclusion Criteria:

* Patients under 18 years of age,
* patients with psychotic disorders with hallucinations and delusions, patients with schizophrenia,
* patients with STAI I-II score below 20 and above 59, patients with PSQI score below 5.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-12-23 (Estimated); Primary Completion 2025-06-02 (Estimated); Study Completion 2025-12-02 (Estimated)

PRIMARY OUTCOMES:
anxiety level -STAI Forms | up to 6 months
  anxiety level, the STAI-II forms

SECONDARY OUTCOMES:
Sleep quality-Pittsburg Sleep Quality Index (PSQI) | up to 6 months
  The Pittsburgh Sleep Quality Index (PSQI)

IPD SHARING:
Plan to Share IPD: No